CLINICAL TRIAL: NCT00460499
Title: Improving Outcomes In Diabetic Patients During CABG Surgery By Optimizing Glycemic Control
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American Heart Association (Other)
Responsible Party: Principal Investigator, Harold L. Lazar MD, Professor of Cardiothoracic Surgery, American Heart Association
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H-23735
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Glycemic Control
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- B Low dose GIK (Active Comparator): This group will have low doses of glucose and insulin
  Interventions: Drug: B Low Dose GIK
- C High Dose GIK (Active Comparator): This group will have high doses of insulin and glucose
  Interventions: Drug: C High Dose GIK
- A Insulin (Active Comparator): This group will receive only an intravenous insulin infusion
  Interventions: Drug: A IV Insulin drip

INTERVENTIONS:
Drug: A IV Insulin drip — These patients will receive 100units of insulin in 100ml of saline intravenously to keep blood glucose between 120-180mg/dl.
  Arms: A Insulin
Drug: B Low Dose GIK — These patients will receive D5W+80unitsInsulin+40mEqKCL IV to keep blood glucose between 120-180mg/dl
  Arms: B Low dose GIK
Drug: C High Dose GIK — This group will receive D20W+160units IV insulin to keep blood sugar between 120-180mg/dl
  Arms: C High Dose GIK

SUMMARY:
This study seeks to determine whether varying the dose of insulin and glucose in diabetic patients during coronary bypass surgery will improve outcomes in these patients.

DETAILED DESCRIPTION:
Our previous study has shown that maintaining serum glucose between 120-180mg/dl in the perioperative period during CABG surgery in diabetic patients improves outcomes. The purpose of this trial is: (1) to determine whether outcomes can be improved by altering the content of glucose or insulin in these solutions (2)to determine the effect of these solutions and glycemic control on the inflammatory response of arterial and venous conduits used during surgery, (3) to determine whether the beneficial effects of improved glycemic control can be correlated with changes in the inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic CABG patients

Exclusion Criteria:

* Renal and hepatic failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2004-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
glycemic control, postoperative morbidity, inflammatory markers | 24 hours following surgery
glycemic control | 24 hours following surgery

SECONDARY OUTCOMES:
free fatty acid levels | 24 hours following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Harold L Lazar MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194
- [Derived] Lazar HL, McDonnell MM, Chipkin S, Fitzgerald C, Bliss C, Cabral H. Effects of aggressive versus moderate glycemic control on clinical outcomes in diabetic coronary artery bypass graft patients. Ann Surg. 2011 Sep;254(3):458-63; discussion 463-4. doi: 10.1097/SLA.0b013e31822c5d78. PMID 21865944